CLINICAL TRIAL: NCT03648632
Title: Stereotactic Radiotherapy (SBRT) in Patients With Locally Advanced Pancreatic Cancer (LAPC). A Danish Phase II Study
Brief Title: Stereotactic Radiotherapy (SBRT) in Patients With Locally Advanced Pancreatic Cancer (LAPC)
Acronym: SBRT-PC-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Per Pfeiffer (Other)
Responsible Party: Sponsor-Investigator, Per Pfeiffer, Professor, MD, PhD, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KFE 18.13
Record Dates: First submitted 2018-06-20; First posted 2018-08-27 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Locally Advanced Pancreatic Cancer
Keywords: Stereotactic Radiotherapy
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Radiotherapy (Experimental): 50 Gy in 5 fractions within a total of 7 - 8 days
  Interventions: Radiation: Stereotactic Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Radiotherapy — Patients should be treated with 50 Gy in 5 fractions within a total of 7 - 8 days.

SUMMARY:
Stereotactic Radiotherapy (SBRT) in patients with locally advanced pancreatic cancer (LAPC).

A Danish phase II study.

DETAILED DESCRIPTION:
Combination chemotherapy (e.g. FOLFIRINOX (5-fluorouracil, irinotecan, oxaliplatin), Gem-Abraxane, Gem-Cap, Gem-S1) is standard of care in patients with LAPC but more and more scientific studies point to the fact that patients without sign of progressive disease (PD) will benefit from additional radiotherapy and especially SBRT.

The sample size is based on Simon's two stages mini-max design. This design ensures early study termination if there is insufficient effect.

A resection rate less than 10% after SBRT is not clinically acceptable. Assuming a significance level at 0.1 (α = 0.1) and a power at 90% (β = 0.10) it can be calculated, that 16 patients should be included in the first part of the study. The enrolment will continue until 16 patients have completed SBRT and have been re-evaluated for resection by CT scan (and endoscopic ultrasonography + laparoscopic ultrasound, if available). If 1 or less out of the first 16 consecutive patients are being resected the investigators will reject our hypotheses and close the study after the first stage of accrual. If 2 or more patients are resected, an additional 9 patients will be accrued in the second stage. If at least 4 out of 25 patients are resected, a true resection rate of 30% cannot be excluded, and the investigators will conclude that the treatment is effective enough to continue with future studies.

To ensure 25 evaluable patients the investigators will include a total of 30 patients.

ELIGIBILITY:
Inclusion Criteria:

* LAPC (Karolinska Type B, C or D1)
* Cytologically or histologically verified adenocarcinoma/carcinoma
* Prior combination chemotherapy for 2-6 months (unless contraindicated) and no sign of progressive disease
* The patient is medically operable (i.e. no co-morbidity which can preclude anaesthesia or surgery)
* World Health Organization performance status 0-1
* Age ≥ 18 years
* Adequate hepatic function: bilirubin <3.0 x Upper Normal Limit, International Normalized Ratio <1.6, Activated Partial Thromboplastin Time < 1,5 x Upper Normal Limit. Patients with obstruction of bile duct or gut must be drained before start of therapy
* Oral and written informed consent must be obtained prior to registration with planned date of first treatment within 14 days from registration.

Exclusion Criteria:

* M1 disease
* Prior radiotherapy to abdominal cavity
* Pregnancy or breast-feeding. Fertile patients must use adequate contraceptives
* Severe uncontrolled concomitant illness (e.g. clinically significant cardiac disease or myocardial infarction within 12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Resection rate for all patients starting SBRT | 12 month
  Resection rate for all patients starting SBRT

SECONDARY OUTCOMES:
1 year survival for all patients starting SBRT | 12 month
  1 year survival for all patients starting SBRT
Progression-free survival (PFS) | 12 month
  PFS will be calculated from the date of registration to the date of documented progressive disease
Overall survival (OS) | 12 month
  OS will be calculated from the date of registration to the date of documented progressive disease
Adverse events grade 2-5 (NCI-CTCAE 4.1) | 12 month
  Adverse events grade 2-5 (NCI-CTCAE 4.1)
Surgical complications, including irreversible electroporation (IRE) (Clavien-Dindo) | 30 days
  Complication rate will be gathered.
Mortality | 30 days
  Mortality rate
Mortality | 90 days
  Mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Per Pfeiffer, Professor, Principal Investigator — Odense Universitetshospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Weisz Ejlsmark M, Bahij R, Schytte T, Ronn Hansen C, Bertelsen A, Mahmood F, Bau Mortensen M, Detlefsen S, Weber B, Bernchou U, Pfeiffer P. Adaptive MRI-guided stereotactic body radiation therapy for locally advanced pancreatic cancer - A phase II study. Radiother Oncol. 2024 Aug;197:110347. doi: 10.1016/j.radonc.2024.110347. Epub 2024 May 28. PMID 38815694